CLINICAL TRIAL: NCT03965208
Title: Safety and Efficacy of Bivalirudin Versus Heparin for Systemic Anticoagulation in Extracorporeal Membrane Oxygenation: an Open Label, Parallel Group Randomized Pilot Study (BIV-ECMO2)
Brief Title: Safety and Efficacy of Bivalirudin Versus Heparin for Systemic Anticoagulation in Extracorporeal Membrane Oxygenation
Acronym: BIV-ECMO2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Legacy Health System (Other)
Collaborators: Pacific University (Other)
Responsible Party: Principal Investigator, R. Brigg Turner, Principal investigator, Legacy Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1665-2019
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Anticoagulants
MeSH Terms: interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Unfractionated heparin (Active Comparator): Patients randomized to this group will receive anticoagulation with unfractionated heparin
  Interventions: Drug: Unfractionated heparin
- Bivalirudin (Experimental): Patients randomized to this group will receive anticoagulation with bivalirudin
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Bivalirudin — titrated continuous infusion
  Other Names: Angiomax
  Arms: Bivalirudin
Drug: Unfractionated heparin — titrated continuous infusion
  Arms: Unfractionated heparin

SUMMARY:
This study will evaluate heparin as compared to bivalirudin for systemic anticoagulation in adult patients that require extracorporeal membrane oxygenation (ECMO). Half of the participants will receive heparin and half will receive bivalirudin.

DETAILED DESCRIPTION:
The investigators will randomly assign 34 adult patients requiring ECMO to receive bivalirudin or unfractionated heparin in a 1:1 fashion. There will be 17 patients in each group for a total of 34 patients.

Unfractionated heparin binds to antithrombin thereby causing an anticoagulant effect while bivalirudin binds directly to thrombin. Use of unfractionated heparin in this population is problematic due to reliance on adequate levels of circulating antithrombin, complex pharmacokinetics, and variable clearance. Bivalirudin avoids many of these difficulties.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Require ECMO and systemic anticoagulation as determined by the primary treating physician
3. Require anticoagulation to target an activated partial thromboplastin time (aPTT) of 40-60 seconds or 60-80 seconds

Exclusion Criteria:

1. Prior inclusion in this study
2. Patients with known or suspected heparin induced thrombocytopenia
3. Systemic anticoagulation at Legacy for ≥ 24 hours during ECMO immediately prior to study enrollment
4. Allergy to heparin or related products or bivalirudin
5. Known anti-thrombin deficiency
6. Selection of a non-standard aPTT target range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in the target anticoagulation range | From ECMO cannulation (start of ECMO) until patient is decannulated up to 12 weeks
  activated partial thromboplastin time

SECONDARY OUTCOMES:
Major bleeding events | From ECMO cannulation (start of ECMO) until patient is decannulated up to 12 weeks
Major clinical thrombotic events | From ECMO cannulation (start of ECMO) until patient is decannulated up to 12 weeks
Duration of oxygenator use | From ECMO cannulation (start of ECMO) until patient is decannulated up to 12 weeks

OTHER OUTCOMES:
Number of blood products received | From ECMO cannulation (start of ECMO) until patient is decannulated up to 12 weeks
Percentage of patients that reach the target anticoagulation range within the first 24 hours | From ECMO cannulation (start of ECMO) until patient is decannulated up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: R Brigg Turner, PharmD, Principal Investigator — Pacific University
Locations (1):
- Legacy Health System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No